CLINICAL TRIAL: NCT01785316
Title: The Scandinavian Randomized Controlled Trial of Isolated Hepatic Perfusion for Uveal Melanoma Liver Metastases
Acronym: SCANDIUM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Karolinska University Hospital (Other); University Hospital, Linkoeping (Other); Uppsala University Hospital (Other); Skane University Hospital (Other); University Hospital, Umeå (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Roger Olofsson Bagge, Associate professor, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SUGBG-013001
Record Dates: First submitted 2013-02-01; First posted 2013-02-07 (Estimated); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Melanoma; Uveal Neoplasms
Keywords: Perfusion Cancer Chemotherapy, Regional
MeSH Terms: conditions — Melanoma; Uveal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IHP (Experimental): Isolated Hepatic Perfusion
  Interventions: Procedure: IHP
- BAC (No Intervention): Best alternative care

INTERVENTIONS:
Procedure: IHP
  Arms: IHP

SUMMARY:
A randomized controlled, open-label, multi-centre study evaluating if Isolated Hepatic Perfusion (IHP) increases Overall Survival compared with Best Alternative Care (BAC) in patients with isolated liver metastases from uveal melanoma.

DETAILED DESCRIPTION:
Uveal melanoma is the most common primary intraocular malignancy in adults. Despite successful control of the primary tumor, metastatic disease will ultimately develop in approximately 50% of the patients. The liver is the most common site for metastases, and about 50% of the patients will have isolated liver metastases. These metastases are generally refractory to systemic chemotherapy and the median survival for patients with liver metastases is about 6 months. Regardless of treatment, the mortality rate is approximately 90% at 2 years with only about 1% of the patients surviving more than 5 years.

Isolated hepatic perfusion (IHP) is a regional treatment that was first performed more than 40 years ago (Aust and Ausman 1960). During IHP, the liver is completely isolated from the systemic circulation, allowing a high concentration of chemotherapy to be perfused through the liver with minimal systemic exposure. In a previous study from our institution, IHP was analysed based on improvements in the procedure and the results showed an improved outcome together with minimized morbidity and mortality over time.

A phase II follow-up study confirms that IHP is a promising technique with tolerable morbidity. There are yet no randomized trials comparing overall survival in IHP, but in an attempt to answer this question the investigators did a register study showing a 14 months increased survival when comparing the patients treated with IHP with the longest surviving patients in Sweden during the same time period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged above 18 years.
2. Signed and dated written informed consent before the start of specific protocol procedures.
3. Histologically or cytologically proven liver metastases of uveal melanoma. If this is not possible at the time of randomization, a biopsy is mandatory before start of treatment.
4. Liver metastases measurable by MRI (preferred) or CT of thorax and abdomen according to RECIST version 1.1 with at least one unidimensional measurable lesion ≥ 10 mm. The examination should be within 4 weeks prior to randomization.
5. ECOG performance status of 0 or 1.
6. No previous chemotherapy, radiotherapy, or biologic therapy for uveal melanoma metastases (ie first-line therapy)
7. Adequate hepatic function (defined as ASAT,ALAT, bilirubin <= 3*ULN and PK-INR <= 1.5) and no medical history of liver cirrhosis or portal hypertension

Exclusion Criteria:

1. More than 50% of the liver volume (measured by CT or MRI) replaced by tumour.
2. Evidence of extrahepatic disease by PET-CT
3. Life expectancy of less than 4 months
4. Pregnant or breast-feeding. Women of childbearing potential must have a negative pregnancy test performed within seven days prior to the start of study.
5. Active infection.
6. Ischemic cardiac disease or history of congestive heart failure with an LVEF < 40%.
7. COPD or other chronic pulmonary disease with PFT's indicating an FEV< 50% predicted for age.
8. Reduced renal function defined as S-Creatinine >=1.5xULN or Creatinine Clearance < 40 mL/min, calculated using the Cockroft and Gault formula.
9. Reduced blood leukocytes or platelets defined as LPK < 2.0x109/L and TPK <100x109/L
10. Use of live vaccines four weeks before or after the start of study.
11. Body mass index above 35.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2013-06-15 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Overall survival | 24 months
  OS defined as the frequency of individuals alive at 24 months

SECONDARY OUTCOMES:
Hepatic progression-free survival | 24 months
  Defined as time from randomization to progress of existing lesions, or appearance of new lesions, within the liver according to RECIST criteria (version 1.1) using CT or MRI.
Response | 24 months
  Defined as best response according to RECIST criteria (version 1.1) using CT or MRI. For the BAC-group, during the whole follow-up of 24 months. For the IHP-group, until hepatic progression (the time point when cross-over to the BAC-group is allowed).
Health economic evaluation | 24 months
  Health economic evaluation measured using QALY calculated using EQ5D-3L at all study visits.
SAE | 24 months
  Number of Participants with SAE as a Measure of Safety

CONTACTS AND LOCATIONS:
Overall Officials: Roger Olofsson Bagge, Dr, Principal Investigator — Department of Surgery, Sahlgrenska University Hospital, Gothenburg, Sweden
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

REFERENCES:
- [Background] Rizell M, Mattson J, Cahlin C, Hafstrom L, Lindner P, Olausson M. Isolated hepatic perfusion for liver metastases of malignant melanoma. Melanoma Res. 2008 Apr;18(2):120-6. doi: 10.1097/CMR.0b013e3282f8e3c9. PMID 18337648
- [Background] Olofsson R, Cahlin C, All-Ericsson C, Hashimi F, Mattsson J, Rizell M, Lindner P. Isolated hepatic perfusion for ocular melanoma metastasis: registry data suggests a survival benefit. Ann Surg Oncol. 2014 Feb;21(2):466-72. doi: 10.1245/s10434-013-3304-z. Epub 2013 Oct 19. PMID 24141377
- [Result] Olofsson Bagge R, Nelson A, Shafazand A, All-Eriksson C, Cahlin C, Elander N, Helgadottir H, Kiilgaard JF, Kinhult S, Ljuslinder I, Mattsson J, Rizell M, Sternby Eilard M, Ullenhag GJ, Nilsson JA, Ny L, Lindner P. Isolated Hepatic Perfusion With Melphalan for Patients With Isolated Uveal Melanoma Liver Metastases: A Multicenter, Randomized, Open-Label, Phase III Trial (the SCANDIUM Trial). J Clin Oncol. 2023 Jun 1;41(16):3042-3050. doi: 10.1200/JCO.22.01705. Epub 2023 Mar 20. PMID 36940407
- [Derived] Olofsson R, Ny L, Eilard MS, Rizell M, Cahlin C, Stierner U, Lonn U, Hansson J, Ljuslinder I, Lundgren L, Ullenhag G, Kiilgaard JF, Nilsson J, Lindner P. Isolated hepatic perfusion as a treatment for uveal melanoma liver metastases (the SCANDIUM trial): study protocol for a randomized controlled trial. Trials. 2014 Aug 9;15:317. doi: 10.1186/1745-6215-15-317. PMID 25106493